CLINICAL TRIAL: NCT07032584
Title: Impact of Multimodal Telerehabilitation on Reducing Disparities in Rural Survivors of Metastatic Prostate Cancer
Brief Title: Impact of Multimodal Telerehabilitation in Rural Patients With Metastatic Prostate Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Huntsman Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HCI177474; HT94252410264 (Other Grant/Funding Number: US DEPARTMENT OF DEFENSE)
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer; Metastatic Prostate Cancer; Androgen Deprivation Therapy
Keywords: Telerehabilitation; Rural Health
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation Intervention (Experimental): Participants in the Telerehabilitation Intervention group (TR) will receive a comprehensive baseline examination conducted by the blinded assessment team. They will also be evaluated by the clinical PT who will prescribe an individualized exercise plan and train them how to perform the exercises. Patients will be mailed exercise equipment (portable bike, elastic bands, pulse oximeter, and activity tracker) with the necessary instructions. Additionally, the TR group will also receive a touchscreen tablet for computer-mediated support in following their individualized exercise plans at their homes daily. The tablet will contain multimedia instructional materials on how to set up and use the telerehab unit.
  Interventions: Other: Telerehabilitation Intervention
- Best Available Care (Other): Participants in the Best Available Care (BAC) group will receive a comprehensive baseline examination conducted by the blinded assessment team. They will also be evaluated by the clinical PT who will prescribe an individualized exercise plan and train them how to perform the exercises. Patients will be mailed exercise equipment (portable bike, elastic bands, pulse oximeter, and activity tracker) with the necessary instructions.
  Interventions: Other: Telerehabilitation Intervention

INTERVENTIONS:
Other: Telerehabilitation Intervention — TheTelerehabilitation Intervention (TR) group utilizes a touchscreen tablet equipped with a computer-guided rehabilitation program that provides ongoing support and feedback for home-based rehabilitation.

SUMMARY:
People with prostate cancer may have a decreased quality of life due to the cancer itself and due to a lifesaving cancer treatment. Physical therapy, including regular exercise, helps patients with cancer to reduce disease symptoms and improve their quality of life. However, cancer rehabilitation programs in rural areas are not readily available and may require constant travel and significant financial resources, which may limit access to these services on a continuous basis.

Technology can allow patients residing in rural areas to exercise at home under the supervision of their rehabilitation team. However, it is unclear how effective this approach is. This research team will conduct a clinical trial in which half of the randomly chosen participants receiving hormonal prostate cancer therapy will use this new technology to exercise at home. Another half - will exercise at home without this new technology. After six months, the study will compare the quality of life and cancer symptoms in these two groups.

The investigators hope that this study will demonstrate that the patients who were helped by the new technology to exercise at home will have better fitness, fewer symptoms, and better quality of life. If the study demonstrates this in this project, other patients with cancer residing in rural areas will be able to take advantage of this technology. This approach can be extended to people with different diseases who have difficulties accessing medical care in rural areas to undergo required physical, cognitive, and occupational rehabilitation, and improve their quality of life.

DETAILED DESCRIPTION:
Background. Prostate cancer patients receiving androgen deprivation therapy frequently experience debilitating side effects significantly affecting their quality of life. Recent studies demonstrated the efficacy of multimodal rehabilitation for secondary and tertiary prevention in prostate cancer patients, reduction of cancer symptoms, and improvements in functional recovery and QOL. Despite the mounting evidence regarding the benefits of multimodal rehabilitation for this population, multiple barriers limit the access of these patients to cancer rehabilitation, especially in rural areas. Telemedicine approaches have the potential to improve access to cancer rehabilitation. This team's previous studies showed a high acceptance of home-based telerehabilitation in older adults with chronic health conditions and cancer and a positive impact on clinical outcomes. In a recent pilot usability study, the investigators demonstrated that multimodal telerehabilitation is well accepted by patients with metastatic bladder cancer who expressed strong interest in home-based cancer telerehabilitation. However, the impact of multimodal telerehabilitation in patients with metastatic prostate cancer residing in rural areas has not been studied systematically. New models to deliver cancer rehabilitation in rural areas are urgently needed.

Objective. The primary objective of the proposed research is to assess the feasibility of an innovative home-based cancer telerehabilitation model in prostate cancer patients undergoing androgen-deprivation therapy by (1) assessing the potential impact of individualized multimodal telerehabilitation on quality of life, fitness, physical activity, and socio-behavioral outcomes; (2) identifying acceptance, needs, and preferences for home telerehabilitation in prostate cancer patients depending on the cancer stage. The proposed multimodal telerehabilitation model allows a rehabilitation therapy team to set up individualized rehabilitation plans using a web-based care management portal and monitor patient progress online. Patients at home follow a safe and effective personalized exercise plan guided by interactive touch-screen technology combined with behavioral counseling, social support, and interactive education. The design of the telerehabilitation system is based on the cloud-based Internet-of-Things architecture allowing real-time monitoring of cardiovascular parameters and exercise performance. The patient's level of exertion during exercise is automatically identified by a validated AI-driven algorithm supporting exercise safety and efficacy.

Primary Aim: (1) Determine the effect of multimodal cancer telerehabilitation on disease-specific quality of life (QoL) in prostate cancer patients receiving androgen deprivation therapy in a pilot randomized controlled trial. The QoL will be the primary endpoint measured by the Functional Assessment of Cancer Therapy-Prostate (FACT-P) scale.

Secondary Aims: (2) Determine the effect of cancer telerehabilitation on the following functional, socio-behavioral, and cognitive outcomes at 6 months: fitness, mobility, exercise self-efficacy, adherence, motivation, cancer symptoms, patient-provider communication, social support, depression, satisfaction with care, and financial toxicity; (3) Identify acceptance, needs, preferences, barriers, and facilitators for home-based cancer telerehabilitation in prostate cancer patients using qualitative analysis; (4) Evaluate primary and secondary aims in specific subgroups stratified by cancer stage and explore possible interactions; (5) Compare the longitudinal trajectories of primary and secondary outcomes in the intervention and control groups. Evaluate relations between primary and secondary outcomes, including quality of life, exercise self-efficacy, adherence, motivation, patient-provider communication, and social support.

Study Design. To evaluate the efficacy of multimodal cancer telerehabilitation, the research team will conduct a randomized clinical trial beginning in month 7 of the project. Seventy-four eligible patients will be enrolled and randomly assigned to one of two study groups: the telerehabilitation (TR) intervention or best available care (BAC) control group. The individual prostate cancer patient receiving ADT and residing in a rural area will be the unit of analysis. For each participant, the study will assess the effect of TR on quality of life, functional outcomes, cancer symptoms, socio-behavioral parameters, financial toxicity, and satisfaction with medical care.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 years or older
2. Confirmed diagnosis of prostate cancer
3. Men receiving standard-of-care ADT either for high-risk, locally advanced prostate cancer or as a part of multicomponent management of metastatic prostate cancer;
4. Residing in a rural community defined by the Rural-Urban Commuting Area (RUCA) codes from the Federal Office of Rural Health Policy (4 and higher).

Exclusion Criteria:

1. Have unstable angina, uncontrolled hypertension, recent myocardial infarction, pacemakers, painful or unstable bony metastases, or recent skeletal fractures.
2. Are engaged in a regular exercise rehabilitation program.
3. Have relocation plans within the next 6 months
4. Participate in another clinical trial related to prostate cancer or rehabilitation. The patients will also be required to have a working telephone line in their home or a cell phone.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy-Prostate (FACT-P) | up to 6 months from baseline
  To assess disease-specific quality of life (QOL) in prostate cancer patients.
  FACT-P is a 5-point Likert scale from "0 Not at all" to "4 Very much". The FACT-P is a 39-item questionnaire with a minimum score of 0 and a maximum score of 156. Lower scores indicate worse QOL, and higher scores indicate better QOL. This outcome measure will report mean FACT-P total score.

SECONDARY OUTCOMES:
30-second Sit-to-Stand Test | up to 6 months from baseline
  To assess functional mobility.
  The 30-second Sit-to-Stand Test records the number of times a participant can come to a full standing position in 30 seconds. This outcome measure will report mean Sit-to-Stand score.
Godin Leisure Score Index | up to 6 months from baseline
  To assess physical activity.
  Godin Leisure Score Index is a questionnaire to assess time spent in leisure exercise. Godin Leisure Score Index is a continuous index, with a minimum of 0. Lower scores indicate lower activity, and higher scores indicate higher activity.
  This outcome measure will report the mean Godin Leisure Score Index.
8-foot Timed Up and Go | up to 6 months from baseline
  To assess functional fitness in study participants.
  The 8-foot Timed Up and Go measures the amount of time participants can stand (from a sitting position), walk 8-feet away, walk 8-feet back, and sit down. This outcome measure will report the mean results in seconds.
FACIT-Fatigue | up to 6 months from baseline
  To assess self-reported fatigue and its impact on daily activities in study participants.
  FACIT-Fatigue is a 5-point Likert scale from "0 Not at all" to "4 Very much". FACIT-Fatigue is a 13-item questionnaire with a minimum score of 0 and a maximum score of 52. Lower scores indicate worse QOL, and higher scores indicate better QOL. This outcome measure will report the mean FACIT-Fatigue total score.
Exercise Self-Efficacy Scale (EXSE) | up to 6 months from baseline
  To assess exercise self-efficacy.
  EXSE assesses exercise self-efficacy, or a patient's belief in their ability to continue regular exercise. This is an 8-item questionnaire. Each item is a 10-point scale, ranging from 0% (NOT AT ALL CONFIDENT) to 100% (Highly CONFIDENT).
  Total score ranges from 0 to 100, with lower scores indicating worse exercise self-efficacy and higher scores indicating better exercise self efficacy.
Behavioral Regulation in Exercise Questionnaire 3 (BREQ-3) | up to 6 months from baseline
  To assess participant exercise motivation.
  BREQ-3 is an assessment measuring a patient's exercise motivation. BREQ-3 reports 6 sub-scores: Amotivation and External, Introjected, Identified, Integrated, and Intrinsic regulation.
  BREQ-3 score ranges from 0 to 96. Lower score means low motivation, higher scores indicate higher motivation
  This outcome measure will report mean BREQ-3.

CONTACTS AND LOCATIONS:
Overall Officials: Manish Kohli, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abetz L, Coombs JH, Keininger DL, Earle CC, Wade C, Bury-Maynard D, Copley-Merriman K, Hsu MA. Development of the cancer therapy satisfaction questionnaire: item generation and content validity testing. Value Health. 2005 Nov-Dec;8 Suppl 1:S41-53. doi: 10.1111/j.1524-4733.2005.00073.x. PMID 16336488
- [Background] National Healthcare Quality and Disparities Report: Chartbook on Rural Healthcare [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2021 Nov. Report No.: 22-0010. Available from http://www.ncbi.nlm.nih.gov/books/NBK576369/ PMID 35263059
- [Background] Akaike H.
- [Background] Alibhai SM, Breunis H, Timilshina N, Johnston C, Tomlinson G, Tannock I, Krahn M, Fleshner NE, Warde P, Canning SD, Klotz L, Naglie G. Impact of androgen-deprivation therapy on physical function and quality of life in men with nonmetastatic prostate cancer. J Clin Oncol. 2010 Dec 1;28(34):5038-45. doi: 10.1200/JCO.2010.29.8091. Epub 2010 Nov 1. PMID 21041715
- [Background] Amireault S, Godin G, Lacombe J, Sabiston CM. The use of the Godin-Shephard Leisure-Time Physical Activity Questionnaire in oncology research: a systematic review. BMC Med Res Methodol. 2015 Aug 12;15:60. doi: 10.1186/s12874-015-0045-7. PMID 26264621
- [Background] Annunziata MA, Muzzatti B, Bidoli E, Flaiban C, Bomben F, Piccinin M, Gipponi KM, Mariutti G, Busato S, Mella S. Hospital Anxiety and Depression Scale (HADS) accuracy in cancer patients. Support Care Cancer. 2020 Aug;28(8):3921-3926. doi: 10.1007/s00520-019-05244-8. Epub 2019 Dec 19. PMID 31858249
- [Background] Basaria S, Lieb J 2nd, Tang AM, DeWeese T, Carducci M, Eisenberger M, Dobs AS. Long-term effects of androgen deprivation therapy in prostate cancer patients. Clin Endocrinol (Oxf). 2002 Jun;56(6):779-86. doi: 10.1046/j.1365-2265.2002.01551.x. PMID 12072048
- [Background] Beck SL, Schwartz AL, Towsley G, Dudley W, Barsevick A. Psychometric evaluation of the Pittsburgh Sleep Quality Index in cancer patients. J Pain Symptom Manage. 2004 Feb;27(2):140-8. doi: 10.1016/j.jpainsymman.2003.12.002. PMID 15157038
- [Background] Bedra M, McNabney M, Stiassny D, Nicholas J, Finkelstein J. Defining patient-centered characteristics of a telerehabilitation system for patients with COPD. Stud Health Technol Inform. 2013;190:24-6. PMID 23823363
- [Background] Bedra M, Finkelstein J. Feasibility of post-acute hip fracture telerehabilitation in older adults. Stud Health Technol Inform. 2015;210:469-73. PMID 25991191
- [Background] Bennett KJ, Pumkam C, Bellinger JD, Probst JC. Cancer screening delivery in persistent poverty rural counties. J Prim Care Community Health. 2011 Oct 1;2(4):240-9. doi: 10.1177/2150131911406123. Epub 2011 May 17. PMID 23804842
- [Background] Benzo R. Satori: Awakening to Outcomes That Matter: The Impact of Social Support in Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2017 Sep;14(9):1385-1386. doi: 10.1513/AnnalsATS.201707-526ED. No abstract available. PMID 28862500
- [Background] Berger AM, Mooney K. Dissemination and Implementation of Guidelines for Cancer-Related Fatigue. J Natl Compr Canc Netw. 2016 Nov;14(11):1336-1338. doi: 10.6004/jnccn.2016.0144. No abstract available. PMID 27799505
- [Background] Blanchard CM, Courneya KS, Rodgers WM, Murnaghan DM. Determinants of exercise intention and behavior in survivors of breast and prostate cancer: an application of the theory of planned behavior. Cancer Nurs. 2002 Apr;25(2):88-95. doi: 10.1097/00002820-200204000-00002. PMID 11984095
- [Background] Bourke L, Sohanpal R, Nanton V, Crank H, Rosario DJ, Saxton JM. A qualitative study evaluating experiences of a lifestyle intervention in men with prostate cancer undergoing androgen suppression therapy. Trials. 2012 Nov 14;13:208. doi: 10.1186/1745-6215-13-208. PMID 23151126
- [Background] Brick R, Padgett L, Jones J, Wood KC, Pergolotti M, Marshall TF, Campbell G, Eilers R, Keshavarzi S, Flores AM, Silver JK, Virani A, Livinski AA, Ahmed MF, Kendig T, Khalid B, Barnett J, Borhani A, Bernard G, Lyons KD. The influence of telehealth-based cancer rehabilitation interventions on disability: a systematic review. J Cancer Surviv. 2023 Dec;17(6):1725-1750. doi: 10.1007/s11764-022-01181-4. Epub 2022 Feb 26. PMID 35218521
- [Background] Brown M, Murphy MH, McAneney H, McBride K, Crawford F, Cole A, O'Sullivan JM, Jain S, Prue G. Feasibility of home-based exercise training during adjuvant treatment for metastatic castrate-resistant prostate cancer patients treated with an androgen receptor pathway inhibitor (EXACT). Support Care Cancer. 2023 Jul 4;31(7):442. doi: 10.1007/s00520-023-07894-1. PMID 37402060
- [Background] Campbell KL, Winters-Stone KM, Wiskemann J, May AM, Schwartz AL, Courneya KS, Zucker DS, Matthews CE, Ligibel JA, Gerber LH, Morris GS, Patel AV, Hue TF, Perna FM, Schmitz KH. Exercise Guidelines for Cancer Survivors: Consensus Statement from International Multidisciplinary Roundtable. Med Sci Sports Exerc. 2019 Nov;51(11):2375-2390. doi: 10.1249/MSS.0000000000002116. PMID 31626055
- [Background] Cella D, Nichol MB, Eton D, Nelson JB, Mulani P. Estimating clinically meaningful changes for the Functional Assessment of Cancer Therapy--Prostate: results from a clinical trial of patients with metastatic hormone-refractory prostate cancer. Value Health. 2009 Jan-Feb;12(1):124-9. doi: 10.1111/j.1524-4733.2008.00409.x. Epub 2008 Jul 18. PMID 18647260
- [Background] Chan ZY, Lim CF, Leow JL, et al. Using the technology acceptance model to examine acceptance of telemedicine by cancer patients in an ambulatory care setting. Proceedings of Singapore Healthcare 2022;31:1-11.
- [Background] Chang P, Zheng J. Updates in Cancer Rehabilitation Telehealth. Curr Phys Med Rehabil Rep. 2022;10(4):332-338. doi: 10.1007/s40141-022-00372-5. Epub 2022 Nov 9. PMID 36408472
- [Background] Cheville AL, Kornblith AB, Basford JR. An examination of the causes for the underutilization of rehabilitation services among people with advanced cancer. Am J Phys Med Rehabil. 2011 May;90(5 Suppl 1):S27-37. doi: 10.1097/PHM.0b013e31820be3be. PMID 21765261
- [Background] Chu D, Popovic M, Chow E, Cella D, Beaumont JL, Lam H, Nguyen J, Di Giovanni J, Pulenzas N, Bedard G, Bottomley A. Development, characteristics and validity of the EORTC QLQ-PR25 and the FACT-P for assessment of quality of life in prostate cancer patients. J Comp Eff Res. 2014 Sep;3(5):523-31. doi: 10.2217/cer.14.41. PMID 25350803
- [Background] Collado L, Brownell I. The crippling financial toxicity of cancer in the United States. Cancer Biol Ther. 2019;20(10):1301-1303. doi: 10.1080/15384047.2019.1632132. Epub 2019 Jul 10. PMID 31291813
- [Background] Cormie P, Galvao DA, Spry N, Joseph D, Taaffe DR, Newton RU. Functional benefits are sustained after a program of supervised resistance exercise in cancer patients with bone metastases: longitudinal results of a pilot study. Support Care Cancer. 2014 Jun;22(6):1537-48. doi: 10.1007/s00520-013-2103-1. Epub 2014 Jan 15. PMID 24424484
- [Background] Crawford-Williams F, Goodwin BC, Chambers SK, Aitken JF, Ford M, Dunn J. Information needs and preferences among rural cancer survivors in Queensland, Australia: a qualitative examination. Aust N Z J Public Health. 2022 Feb;46(1):81-86. doi: 10.1111/1753-6405.13163. Epub 2021 Nov 11. PMID 34761849
- [Background] Cross RK, Cheevers N, Rustgi A, Langenberg P, Finkelstein J. Randomized, controlled trial of home telemanagement in patients with ulcerative colitis (UC HAT). Inflamm Bowel Dis. 2012 Jun;18(6):1018-25. doi: 10.1002/ibd.21795. Epub 2011 Jun 17. PMID 21688350
- [Background] Damschroder LJ, Aron DC, Keith RE, Kirsh SR, Alexander JA, Lowery JC. Fostering implementation of health services research findings into practice: a consolidated framework for advancing implementation science. Implement Sci. 2009 Aug 7;4:50. doi: 10.1186/1748-5908-4-50. PMID 19664226
- [Background] Damschroder LJ, Reardon CM, Widerquist MAO, Lowery J. The updated Consolidated Framework for Implementation Research based on user feedback. Implement Sci. 2022 Oct 29;17(1):75. doi: 10.1186/s13012-022-01245-0. PMID 36309746
- [Background] DiBlasio CJ, Hammett J, Malcolm JB, Judge BA, Womack JH, Kincade MC, Ogles ML, Mancini JG, Patterson AL, Wake RW, Derweesh IH. Prevalence and predictive factors for the development of de novo psychiatric illness in patients receiving androgen deprivation therapy for prostate cancer. Can J Urol. 2008 Oct;15(5):4249-56; discussion 4256. PMID 18814813
- [Background] Dacal K, Sereika SM, Greenspan SL. Quality of life in prostate cancer patients taking androgen deprivation therapy. J Am Geriatr Soc. 2006 Jan;54(1):85-90. doi: 10.1111/j.1532-5415.2005.00567.x. PMID 16420202
- [Background] Drouin H, Walker J, McNeil H, Elliott J, Stolee P. Measured outcomes of chronic care programs for older adults: a systematic review. BMC Geriatr. 2015 Oct 26;15:139. doi: 10.1186/s12877-015-0136-7. PMID 26503159
- [Background] Eaves YD. A synthesis technique for grounded theory data analysis. J Adv Nurs. 2001 Sep;35(5):654-63. doi: 10.1046/j.1365-2648.2001.01897.x. PMID 11529967
- [Background] Edward J, Petermann VM, Eberth JM, Zahnd WE, Vanderpool RC, Askelson N, Rohweder CL, Gonzalez SK, Stradtman LR, Ko LK, Farris PE. Interventions to address cancer-related financial toxicity: Recommendations from the field. J Rural Health. 2022 Sep;38(4):817-826. doi: 10.1111/jrh.12637. Epub 2021 Dec 3. PMID 34861066
- [Background] Elliott J, Fallows A, Staetsky L, Smith PW, Foster CL, Maher EJ, Corner J. The health and well-being of cancer survivors in the UK: findings from a population-based survey. Br J Cancer. 2011 Nov 8;105 Suppl 1(Suppl 1):S11-20. doi: 10.1038/bjc.2011.418. PMID 22048028
- [Background] Evans HE, Forbes CC, Galvao DA, Vandelanotte C, Newton RU, Wittert G, Chambers S, Vincent AD, Kichenadasse G, Girard D, Brook N, Short CE. Usability, Acceptability, and Safety Analysis of a Computer-Tailored Web-Based Exercise Intervention (ExerciseGuide) for Individuals With Metastatic Prostate Cancer: Multi-Methods Laboratory-Based Study. JMIR Cancer. 2021 Jul 28;7(3):e28370. doi: 10.2196/28370. PMID 34318759
- [Background] Evans HEL, Galvao DA, Forbes CC, Girard D, Vandelanotte C, Newton RU, Vincent AD, Wittert G, Kichenadasse G, Chambers S, Brook N, Short CE. Acceptability and Preliminary Efficacy of a Web- and Telephone-Based Personalised Exercise Intervention for Individuals with Metastatic Prostate Cancer: The ExerciseGuide Pilot Randomised Controlled Trial. Cancers (Basel). 2021 Nov 25;13(23):5925. doi: 10.3390/cancers13235925. PMID 34885036
- [Background] Esper P, Mo F, Chodak G, Sinner M, Cella D, Pienta KJ. Measuring quality of life in men with prostate cancer using the functional assessment of cancer therapy-prostate instrument. Urology. 1997 Dec;50(6):920-8. doi: 10.1016/S0090-4295(97)00459-7. PMID 9426724
- [Background] Figueiredo PHS, Veloso LRS, Lima MMO, Vieira CFD, Alves FL, Lacerda ACR, Lima VP, Rodrigues VGB, Maciel EHB, Costa HS. The reliability and validity of the 30-seconds sit-to-stand test and its capacity for assessment of the functional status of hemodialysis patients. J Bodyw Mov Ther. 2021 Jul;27:157-164. doi: 10.1016/j.jbmt.2021.02.020. Epub 2021 Mar 4. PMID 34391227
- [Background] Finkelstein J, Cabrera MR, Hripcsak G. Internet-based home asthma telemonitoring: can patients handle the technology? Chest. 2000 Jan;117(1):148-55. doi: 10.1378/chest.117.1.148. PMID 10631213
- [Background] Finkelstein J, Amelung P. Quality of Life in Asthma Patients is Affected by Home Telemanagement. Value in Health 2005;8(3):246.
- [Background] Finkelstein J, Lapshin O. Reducing depression stigma using a web-based program. Int J Med Inform. 2007 Oct;76(10):726-34. doi: 10.1016/j.ijmedinf.2006.07.004. Epub 2006 Sep 20. PMID 16996299
- [Background] Finkelstein J, Lapshin O, Wasserman E. Randomized study of different anti-stigma media. Patient Educ Couns. 2008 May;71(2):204-14. doi: 10.1016/j.pec.2008.01.002. Epub 2008 Mar 4. PMID 18289823
- [Background] Finkelstein J, Lapshin O, Castro H, Cha E, Provance PG. Home-based physical telerehabilitation in patients with multiple sclerosis: a pilot study. J Rehabil Res Dev. 2008;45(9):1361-73. PMID 19319760
- [Background] Finkelstein J, Lapshin O, Cha E. Feasibility of promoting smoking cessation among methadone users using multimedia computer-assisted education. J Med Internet Res. 2008 Nov 3;10(5):e33. doi: 10.2196/jmir.1089. PMID 18984556
- [Background] Finkelstein J, Cha E. Hypertension telemanagement in blacks. Circ Cardiovasc Qual Outcomes. 2009 May;2(3):272-8. doi: 10.1161/CIRCOUTCOMES.109.849968. PMID 20031848
- [Background] Finkelstein J, Wood J, Cha E. Impact of physical telerehabilitation on functional outcomes in seniors with mobility limitations. Annu Int Conf IEEE Eng Med Biol Soc. 2012;2012:5827-32. doi: 10.1109/EMBC.2012.6347319. PMID 23367254
- [Background] Finkelstein J, Cha E, Dennison CR. Exploring feasibility of home telemanagement in African Americans with congestive heart failure. Stud Health Technol Inform. 2010;160(Pt 1):535-9. PMID 20841744
- [Background] Finkelstein J, Wood J. Using individualized continuous patient education (iCOPE) platform to facilitate smoking cessation in hospitalized patients. Proc. of the 2012 International Symposium on Information Technology in Medicine and Education (ITME), 2012(Vol. 2):727-731.
- [Background] Finkelstein J, Knight A, Marinopoulos S, Gibbons MC, Berger Z, Aboumatar H, Wilson RF, Lau BD, Sharma R, Bass EB. Enabling patient-centered care through health information technology. Evid Rep Technol Assess (Full Rep). 2012 Jun;(206):1-1531. PMID 24422882
- [Background] Finkelstein J, Cha E, Wood J, Wallin MT. Predictors of successful acceptance of home telemanagement in veterans with Multiple Sclerosis. Annu Int Conf IEEE Eng Med Biol Soc. 2013;2013:7314-7. doi: 10.1109/EMBC.2013.6611247. PMID 24111434
- [Background] Finkelstein J, Jeong Ic. Remotely controlled cycling exercise system for home-based telerehabilitation. Annu Int Conf IEEE Eng Med Biol Soc. 2013;2013:7310-3. doi: 10.1109/EMBC.2013.6611246. PMID 24111433
- [Background] Finkelstein J, Jeong IC. Design and Implementation of Home Automated Telemanagement Platform for Interactive Biking Exercise (iBikE HAT). Proc. of the IEEE-EMBS Special Topic Conference on Point-of-Care Healthcare Technologies (POCHT2013), 2013, pp. 236-239.
- [Background] Finkelstein J, Cha E, Royal W. Predictors of Acceptance of Using Games for Cognitive Rehabilitation. Int J of MS Care 2013;15(Suppl 3):35.
- [Background] Finkelstein J, Bedra M. Avatar-based Interactive Diabetes Education in Older Adults. Journal of the American Geriatrics Society 2015;62:S64.
- [Background] Finkelstein J, Bedra M, Li X, Wood J, Ouyang P. Mobile App to Reduce Inactivity in Sedentary Overweight Women. Stud Health Technol Inform. 2015;216:89-92. PMID 26262016
- [Background] Finkelstein J, Cha EM. Using a Mobile App to Promote Smoking Cessation in Hospitalized Patients. JMIR Mhealth Uhealth. 2016 May 6;4(2):e59. doi: 10.2196/mhealth.5149. PMID 27154792
- [Background] Finkelstein J, Wood J, Crew KD, Kukafka R. Introducing a Comprehensive Informatics Framework to Promote Breast Cancer Risk Assessment and Chemoprevention in the Primary Care Setting. AMIA Jt Summits Transl Sci Proc. 2017 Jul 26;2017:58-67. eCollection 2017. PMID 28815107
- [Background] Finkelstein J, Robins D, Liu J. Usability Inspection of Multipurpose Scalable Informed Consent Platform. Stud Health Technol Inform. 2019 Jul 4;262:198-201. doi: 10.3233/SHTI190052. PMID 31349301
- [Background] Finkelstein J, Jeong IC, Doerstling M, Shen Y, Wei C, Karpatkin H. Usability of Remote Assessment of Exercise Capacity for Pulmonary Telerehabilitation Program. Stud Health Technol Inform. 2020 Nov 23;275:72-76. doi: 10.3233/SHTI200697. PMID 33227743
- [Background] Finkelstein J, Huo X, Parvanova I, Galsky M. Usability Inspection of a Mobile Cancer Telerehabilitation System. Stud Health Technol Inform. 2022 Jan 14;289:405-409. doi: 10.3233/SHTI210944. PMID 35062177
- [Background] Finkelstein J, Parvanova I, Huo X. Feasibility of a Virtual Reality App to Promote Pulmonary Rehabilitation. Stud Health Technol Inform. 2023 May 18;302:458-462. doi: 10.3233/SHTI230172. PMID 37203716
- [Background] Fleg JL, Keteyian SJ, Peterson PN, Benzo R, Finkelstein J, Forman DE, Gaalema DE, Cooper LS, Punturieri A, Joseph L, Shero S, Zieman S. Increasing Use of Cardiac and Pulmonary Rehabilitation in Traditional and Community Settings: OPPORTUNITIES TO REDUCE HEALTH CARE DISPARITIES. J Cardiopulm Rehabil Prev. 2020 Nov;40(6):350-355. doi: 10.1097/HCR.0000000000000527. PMID 33074849
- [Background] Gabriel AS, Tsai TY, Xhakli T, Finkelstein J. Patient Perceptions of a Virtual Reality-Based System for Pulmonary Rehabilitation: A Qualitative Analysis. Stud Health Technol Inform. 2023 Jun 29;305:406-409. doi: 10.3233/SHTI230517. PMID 37387051
- [Background] Gabriel AS, Parvanova I, Tsai TY, Finkelstein J. Assessing Patient Perspectives of a Cancer Telerehabilitation Platform Using Thematic Analysis of Semi-Structured Qualitative Interviews. AMIA Jt Summits Transl Sci Proc. 2023 Jun 16;2023:216-224. eCollection 2023. PMID 37350908
- [Background] Gell NM, Dittus K, Caefer J, Martin A, Bae M, Patel KV. Remotely delivered exercise to older rural cancer survivors: a randomized controlled pilot trial. J Cancer Surviv. 2024 Apr;18(2):596-605. doi: 10.1007/s11764-022-01292-y. Epub 2022 Nov 14. PMID 36374436
- [Background] Gerteis M, Edgman-Levitan S, Daley J, Delbanco TL Through the Patient's Eyes: Understanding and Promoting Patient-Centered Care. San Francisco, CA: Jossey-Bass; 1993.
- [Background] Gomez CA, Kleinman DV, Pronk N, Wrenn Gordon GL, Ochiai E, Blakey C, Johnson A, Brewer KH. Addressing Health Equity and Social Determinants of Health Through Healthy People 2030. J Public Health Manag Pract. 2021 Nov-Dec 01;27(Suppl 6):S249-S257. doi: 10.1097/PHH.0000000000001297. PMID 33729197
- [Background] Graves KD. Social cognitive theory and cancer patients' quality of life: a meta-analysis of psychosocial intervention components. Health Psychol. 2003 Mar;22(2):210-9. PMID 12683741
- [Background] Grover A, Joshi A. An overview of chronic disease models: a systematic literature review. Glob J Health Sci. 2014 Oct 29;7(2):210-27. doi: 10.5539/gjhs.v7n2p210. PMID 25716407
- [Background] Harris Insights & Analytics. ASCO 2018 Cancer Opinions Survey, 2018.
- [Background] Hart NH, Poprawski DM, Ashbury F, Fitch MI, Chan RJ, Newton RU, Campbell KL. Exercise for people with bone metastases: MASCC endorsed clinical recommendations developed by the International Bone Metastases Exercise Working Group. Support Care Cancer. 2022 Sep;30(9):7061-7065. doi: 10.1007/s00520-022-07212-1. No abstract available. PMID 35710641
- [Background] Hashibe M, Kirchhoff AC, Kepka D, Kim J, Millar M, Sweeney C, Herget K, Monroe M, Henry NL, Lopez AM, Mooney K. Disparities in cancer survival and incidence by metropolitan versus rural residence in Utah. Cancer Med. 2018 Apr;7(4):1490-1497. doi: 10.1002/cam4.1382. Epub 2018 Mar 13. PMID 29533005
- [Background] Hays RD, Kravitz RL, Mazel RM, Sherbourne CD, DiMatteo MR, Rogers WH, Greenfield S. The impact of patient adherence on health outcomes for patients with chronic disease in the Medical Outcomes Study. J Behav Med. 1994 Aug;17(4):347-60. doi: 10.1007/BF01858007. PMID 7966257
- [Background] Hirko KA, Xu H, Rogers LQ, Martin MY, Roy S, Kelly KM, Christy SM, Ashing KT, Yi JC, Lewis-Thames MW, Meade CD, Lu Q, Gwede CK, Nemeth J, Ceballos RM, Menon U, Cueva K, Yeary K, Klesges LM, Baskin ML, Alcaraz KI, Ford S. Cancer disparities in the context of rurality: risk factors and screening across various U.S. rural classification codes. Cancer Causes Control. 2022 Aug;33(8):1095-1105. doi: 10.1007/s10552-022-01599-2. Epub 2022 Jun 30. PMID 35773504
- [Background] Hussain M, Tangen CM, Berry DL, Higano CS, Crawford ED, Liu G, Wilding G, Prescott S, Kanaga Sundaram S, Small EJ, Dawson NA, Donnelly BJ, Venner PM, Vaishampayan UN, Schellhammer PF, Quinn DI, Raghavan D, Ely B, Moinpour CM, Vogelzang NJ, Thompson IM Jr. Intermittent versus continuous androgen deprivation in prostate cancer. N Engl J Med. 2013 Apr 4;368(14):1314-25. doi: 10.1056/NEJMoa1212299. PMID 23550669
- [Background] Jackson DN, Trivedi N, Baur C. Re-Prioritizing Digital Health and Health Literacy in Healthy People 2030 to Affect Health Equity. Health Commun. 2021 Sep;36(10):1155-1162. doi: 10.1080/10410236.2020.1748828. Epub 2020 Apr 30. PMID 32354233
- [Background] Jeong IC, Karpatkin H, Finkelstein J. Physical Telerehabilitation Improves Quality of Life in Patients with Multiple Sclerosis. Stud Health Technol Inform. 2021 Dec 15;284:384-388. doi: 10.3233/SHTI210752. PMID 34920553
- [Background] Joyce DD, Wallis CJD, Huang LC, Hoffman KE, Zhao Z, Koyama T, Goodman M, Hamilton AS, Wu XC, Paddock LE, Stroup A, Cooperberg MR, Hashibe M, O'Neil BB, Kaplan SH, Greenfield S, Penson DF, Barocas DA. The Association Between Financial Toxicity and Treatment Regret in Men With Localized Prostate Cancer. JNCI Cancer Spectr. 2022 Nov 1;6(6):pkac071. doi: 10.1093/jncics/pkac071. PMID 36255249
- [Background] Kamal SA, Shafiq M and Kakria P. Investigating acceptance of telemedicine services through an extended technology acceptance model (TAM). Technol Soc 2020; 60: 101212.
- [Background] Kang DW, Boule NG, Field CJ, Fairey AS, Courneya KS. Effects of supervised high-intensity interval training on motivational outcomes in men with prostate cancer undergoing active surveillance: results from a randomized controlled trial. Int J Behav Nutr Phys Act. 2022 Sep 29;19(1):126. doi: 10.1186/s12966-022-01365-2. PMID 36175907
- [Background] Khan HM, Ramsey S, Shankaran V. Financial Toxicity in Cancer Care: Implications for Clinical Care and Potential Practice Solutions. J Clin Oncol. 2023 Jun 1;41(16):3051-3058. doi: 10.1200/JCO.22.01799. Epub 2023 Apr 18. PMID 37071839
- [Background] Kirk MA, Kelley C, Yankey N, Birken SA, Abadie B, Damschroder L. A systematic review of the use of the Consolidated Framework for Implementation Research. Implement Sci. 2016 May 17;11:72. doi: 10.1186/s13012-016-0437-z. PMID 27189233
- [Background] Konijeti R, Kibel AS. Androgen deprivation therapy for localized and nonmetastatic prostate cancer: too much of a good thing? Eur Urol. 2012 Jun;61(6):1129-30; discussion 1131. doi: 10.1016/j.eururo.2012.03.002. Epub 2012 Mar 13. No abstract available. PMID 22445550
- [Background] Langlais CS, Chen YH, Van Blarigan EL, Chan JM, Ryan CJ, Zhang L, Borno HT, Newton RU, Luke A, Bang AS, Panchal N, Tenggara I, Schultz B, Lavaki E, Pinto N, Aggarwal R, Friedlander T, Koshkin VS, Harzstark AL, Small EJ, Kenfield SA. Quality of life for men with metastatic castrate-resistant prostate cancer participating in an aerobic and resistance exercise pilot intervention. Urol Oncol. 2023 Mar;41(3):146.e1-146.e11. doi: 10.1016/j.urolonc.2022.11.016. Epub 2022 Dec 15. PMID 36528473
- [Background] Lentz R, Benson AB 3rd, Kircher S. Financial toxicity in cancer care: Prevalence, causes, consequences, and reduction strategies. J Surg Oncol. 2019 Jul;120(1):85-92. doi: 10.1002/jso.25374. Epub 2019 Jan 16. PMID 30650186
- [Background] Levine RL. Healthy People 2030: A Beacon for Addressing Health Disparities and Health Equity. J Public Health Manag Pract. 2021 Nov-Dec 01;27(Suppl 6):S220-S221. doi: 10.1097/PHH.0000000000001409. No abstract available. PMID 34559739
- [Background] Lewis-Thames MW, Langston ME, Khan S, Han Y, Fuzzell L, Xu S, Moore JX. Racial and Ethnic Differences in Rural-Urban Trends in 5-Year Survival of Patients With Lung, Prostate, Breast, and Colorectal Cancers: 1975-2011 Surveillance, Epidemiology, and End Results (SEER). JAMA Netw Open. 2022 May 2;5(5):e2212246. doi: 10.1001/jamanetworkopen.2022.12246. PMID 35587350
- [Background] Lin CC, Bruinooge SS, Kirkwood MK, Olsen C, Jemal A, Bajorin D, Giordano SH, Goldstein M, Guadagnolo BA, Kosty M, Hopkins S, Yu JB, Arnone A, Hanley A, Stevens S, Hershman DL. Association Between Geographic Access to Cancer Care, Insurance, and Receipt of Chemotherapy: Geographic Distribution of Oncologists and Travel Distance. J Clin Oncol. 2015 Oct 1;33(28):3177-85. doi: 10.1200/JCO.2015.61.1558. Epub 2015 Aug 24. PMID 26304878
- [Background] Litwin MS, Tan HJ. The Diagnosis and Treatment of Prostate Cancer: A Review. JAMA. 2017 Jun 27;317(24):2532-2542. doi: 10.1001/jama.2017.7248. PMID 28655021
- [Background] Langley RE, Gilbert DC, Duong T, Clarke NW, Nankivell M, Rosen SD, Mangar S, Macnair A, Sundaram SK, Laniado ME, Dixit S, Madaan S, Manetta C, Pope A, Scrase CD, Mckay S, Muazzam IA, Collins GN, Worlding J, Williams ST, Paez E, Robinson A, McFarlane J, Deighan JV, Marshall J, Forcat S, Weiss M, Kockelbergh R, Alhasso A, Kynaston H, Parmar M. Transdermal oestradiol for androgen suppression in prostate cancer: long-term cardiovascular outcomes from the randomised Prostate Adenocarcinoma Transcutaneous Hormone (PATCH) trial programme. Lancet. 2021 Feb 13;397(10274):581-591. doi: 10.1016/S0140-6736(21)00100-8. PMID 33581820
- [Background] Levine GN, D'Amico AV, Berger P, Clark PE, Eckel RH, Keating NL, Milani RV, Sagalowsky AI, Smith MR, Zakai N; American Heart Association Council on Clinical Cardiology and Council on Epidemiology and Prevention, the American Cancer Society, and the American Urological Association. Androgen-deprivation therapy in prostate cancer and cardiovascular risk: a science advisory from the American Heart Association, American Cancer Society, and American Urological Association: endorsed by the American Society for Radiation Oncology. CA Cancer J Clin. 2010 May-Jun;60(3):194-201. doi: 10.3322/caac.20061. Epub 2010 Feb 2. No abstract available. PMID 20124400
- [Background] Magnan S, Zarychanski R, Pilote L, Bernier L, Shemilt M, Vigneault E, Fradet V, Turgeon AF. Intermittent vs Continuous Androgen Deprivation Therapy for Prostate Cancer: A Systematic Review and Meta-analysis. JAMA Oncol. 2015 Dec;1(9):1261-9. doi: 10.1001/jamaoncol.2015.2895. PMID 26378418
- [Background] Markland D, Tobin V. A modification to the behavioural regulation in exercise questionnaire to include an assessment of amotivation. Journal of Sport and Exercise Psychology. 2004 Jun 1;26(2):191-6.
- [Background] Morris BB, Rossi B, Fuemmeler B. The role of digital health technology in rural cancer care delivery: A systematic review. J Rural Health. 2022 Jun;38(3):493-511. doi: 10.1111/jrh.12619. Epub 2021 Sep 4. PMID 34480506
- [Background] Michie S, van Stralen MM, West R. The behaviour change wheel: a new method for characterising and designing behaviour change interventions. Implement Sci. 2011 Apr 23;6:42. doi: 10.1186/1748-5908-6-42. PMID 21513547
- [Background] Monga U, Garber SL, Thornby J, Vallbona C, Kerrigan AJ, Monga TN, Zimmermann KP. Exercise prevents fatigue and improves quality of life in prostate cancer patients undergoing radiotherapy. Arch Phys Med Rehabil. 2007 Nov;88(11):1416-22. doi: 10.1016/j.apmr.2007.08.110. PMID 17964881
- [Background] Nielsen S, O'Neil B, Chang CP, Mark B, Snyder J, Deshmukh V, Newman M, Date A, Galvao C, Henry NL, Lloyd S, Hashibe M. Determining the association of rurality and cardiovascular disease among prostate cancer survivors. Urol Oncol. 2023 Oct;41(10):429.e15-429.e23. doi: 10.1016/j.urolonc.2023.06.008. Epub 2023 Jul 16. PMID 37455231
- [Background] Northouse L, Schafenacker A, Barr KL, Katapodi M, Yoon H, Brittain K, Song L, Ronis DL, An L. A tailored Web-based psychoeducational intervention for cancer patients and their family caregivers. Cancer Nurs. 2014 Sep-Oct;37(5):321-30. doi: 10.1097/NCC.0000000000000159. PMID 24945270
- [Background] Pagliarulo V, Bracarda S, Eisenberger MA, Mottet N, Schroder FH, Sternberg CN, Studer UE. Contemporary role of androgen deprivation therapy for prostate cancer. Eur Urol. 2012 Jan;61(1):11-25. doi: 10.1016/j.eururo.2011.08.026. Epub 2011 Aug 19. PMID 21871711
- [Background] Park J, Rho MJ, Moon HW, Park YH, Kim CS, Jeon SS, Kang M, Lee JY. Prostate cancer trajectory-map: clinical decision support system for prognosis management of radical prostatectomy. Prostate Int. 2021 Mar;9(1):25-30. doi: 10.1016/j.prnil.2020.06.003. Epub 2020 Jul 30. PMID 33912511
- [Background] Pasek M, Suchocka L, Gasior K. Model of Social Support for Patients Treated for Cancer. Cancers (Basel). 2021 Sep 24;13(19):4786. doi: 10.3390/cancers13194786. PMID 34638270
- [Background] Patel KB, Turner K, Alishahi Tabriz A, Gonzalez BD, Oswald LB, Nguyen OT, Hong YR, Jim HSL, Nichols AC, Wang X, Robinson E, Naso C, Spiess PE. Estimated Indirect Cost Savings of Using Telehealth Among Nonelderly Patients With Cancer. JAMA Netw Open. 2023 Jan 3;6(1):e2250211. doi: 10.1001/jamanetworkopen.2022.50211. PMID 36626174
- [Background] Patrick K, Intille SS, Zabinski MF. An ecological framework for cancer communication: implications for research. J Med Internet Res. 2005 Jul 1;7(3):e23. doi: 10.2196/jmir.7.3.e23. PMID 15998614
- [Background] Pergolotti M, Deal AM, Lavery J, Reeve BB, Muss HB. The prevalence of potentially modifiable functional deficits and the subsequent use of occupational and physical therapy by older adults with cancer. J Geriatr Oncol. 2015 May;6(3):194-201. doi: 10.1016/j.jgo.2015.01.004. Epub 2015 Jan 19. PMID 25614296
- [Background] Plotnikoff R, Blanchard C, Hotz S, Rhodes R. Validation of the decisional balance constructs of the transtheoretical model in the exercise domain: A longitudinal test in a population sample. Measurement in Physical Education and Exercise Science 2001;5(4):191-206.
- [Background] Raedeke TD, Dlugonski D. High Versus Low Theoretical Fidelity Pedometer Intervention Using Social-Cognitive Theory on Steps and Self-Efficacy. Res Q Exerc Sport. 2017 Dec;88(4):436-446. doi: 10.1080/02701367.2017.1368976. Epub 2017 Sep 20. PMID 28929950
- [Background] Rammant E, Bultijnck R, Caperchione CM, Trinh L; research collaboration group of the cancer prevention and management Special Interest Group of ISBNPA. The Use of Theory to Develop Physical Activity Interventions in Urological Cancer Survivors: A Narrative Review. Semin Oncol Nurs. 2021 Feb;37(1):151109. doi: 10.1016/j.soncn.2020.151109. Epub 2021 Jan 28. PMID 33516584
- [Background] Ratcliff R, Voskuilen C, McKoon G. Internal and external sources of variability in perceptual decision-making. Psychol Rev. 2018 Jan;125(1):33-46. doi: 10.1037/rev0000080. Epub 2017 Oct 16. PMID 29035076
- [Background] Rawla P. Epidemiology of Prostate Cancer. World J Oncol. 2019 Apr;10(2):63-89. doi: 10.14740/wjon1191. Epub 2019 Apr 20. PMID 31068988
- [Background] Reddy S, Bruera E, Pace E, Zhang K, Reyes-Gibby CC. Clinically important improvement in the intensity of fatigue in patients with advanced cancer. J Palliat Med. 2007 Oct;10(5):1068-75. doi: 10.1089/jpm.2007.0007. PMID 17985963
- [Background] Resnick B, Zimmerman SI, Orwig D, Furstenberg AL, Magaziner J. Outcome expectations for exercise scale: utility and psychometrics. J Gerontol B Psychol Sci Soc Sci. 2000 Nov;55(6):S352-6. doi: 10.1093/geronb/55.6.s352. PMID 11078112
- [Background] Robins D, Brody R, Jeong IC, Parvanova I, Liu J, Finkelstein J. Towards a Highly Usable, Mobile Electronic Platform for Patient Recruitment and Consent Management. Stud Health Technol Inform. 2020 Jun 16;270:1066-1070. doi: 10.3233/SHTI200325. PMID 32570545
- [Background] Robins D, Brody R, Parvanova I, Finkelstein J. Cognitive Testing of an Electronic Consent Platform: Researcher Perspectives. Stud Health Technol Inform. 2021 Dec 15;284:457-462. doi: 10.3233/SHTI210772. PMID 34920571
- [Background] Rocco P, Finkelstein J. Telerehabilitation for Patients with Cancer: A Scoping Review. Stud Health Technol Inform. 2022 Jun 6;290:543-546. doi: 10.3233/SHTI220136. PMID 35673075
- [Background] Rolenz E, Reneker JC. Validity of the 8-Foot Up and Go, Timed Up and Go, and Activities-Specific Balance Confidence Scale in older adults with and without cognitive impairment. J Rehabil Res Dev. 2016;53(4):511-8. doi: 10.1682/JRRD.2015.03.0042. PMID 27532337
- [Background] Ross J, Stevenson F, Lau R, Murray E. Factors that influence the implementation of e-health: a systematic review of systematic reviews (an update). Implement Sci. 2016 Oct 26;11(1):146. doi: 10.1186/s13012-016-0510-7. PMID 27782832
- [Background] Rubin DB. Multiple imputation after 18+ years (with discussion). Journal of the American Statistical Association 1996;91:473-489.
- [Background] Moses KA, Sprenkle PC, Bahler C, Box G, Carlsson SV, Catalona WJ, Dahl DM, Dall'Era M, Davis JW, Drake BF, Epstein JI, Etzioni RB, Farrington TA, Garraway IP, Jarrard D, Kauffman E, Kaye D, Kibel AS, LaGrange CA, Maroni P, Ponsky L, Reys B, Salami SS, Sanchez A, Seibert TM, Shaneyfelt TM, Smaldone MC, Sonn G, Tyson MD, Vapiwala N, Wake R, Washington S, Yu A, Yuh B, Berardi RA, Freedman-Cass DA. NCCN Guidelines(R) Insights: Prostate Cancer Early Detection, Version 1.2023. J Natl Compr Canc Netw. 2023 Mar;21(3):236-246. doi: 10.6004/jnccn.2023.0014. PMID 36898362
- [Background] Schroder FH, Kurth KH, Fossa SD, Hoekstra W, Karthaus PP, De Prijck L, Collette L. Early versus delayed endocrine treatment of T2-T3 pN1-3 M0 prostate cancer without local treatment of the primary tumour: final results of European Organisation for the Research and Treatment of Cancer protocol 30846 after 13 years of follow-up (a randomised controlled trial). Eur Urol. 2009 Jan;55(1):14-22. doi: 10.1016/j.eururo.2008.09.008. Epub 2008 Sep 17. PMID 18823693
- [Background] Settle JR, Maloni HW, Bedra M, Finkelstein J, Zhan M, Wallin MT. Monitoring medication adherence in multiple sclerosis using a novel web-based tool: A pilot study. J Telemed Telecare. 2016 Jun;22(4):225-33. doi: 10.1177/1357633X15597115. Epub 2015 Aug 6. PMID 26253748
- [Background] Skrabal Ross X, Gunn KM, Olver I. Understanding the strategies rural cancer patients and survivors use to manage financial toxicity and the broader implications on their lives. Support Care Cancer. 2021 Sep;29(9):5487-5496. doi: 10.1007/s00520-021-06086-z. Epub 2021 Mar 12. PMID 33710410
- [Background] Segal RJ, Reid RD, Courneya KS, Malone SC, Parliament MB, Scott CG, Venner PM, Quinney HA, Jones LW, D'Angelo ME, Wells GA. Resistance exercise in men receiving androgen deprivation therapy for prostate cancer. J Clin Oncol. 2003 May 1;21(9):1653-9. doi: 10.1200/JCO.2003.09.534. PMID 12721238
- [Background] Segal RJ, Reid RD, Courneya KS, Sigal RJ, Kenny GP, Prud'Homme DG, Malone SC, Wells GA, Scott CG, Slovinec D'Angelo ME. Randomized controlled trial of resistance or aerobic exercise in men receiving radiation therapy for prostate cancer. J Clin Oncol. 2009 Jan 20;27(3):344-51. doi: 10.1200/JCO.2007.15.4963. Epub 2008 Dec 8. PMID 19064985
- [Background] Sheill G, Brady L, Hayes B, Baird AM, Guinan E, Vishwakarma R, Brophy C, Vlajnic T, Casey O, Murphy V, Greene J, Allott E, Hussey J, Cahill F, Van Hemelrijck M, Peat N, Mucci L, Cunningham M, Grogan L, Lynch T, Manecksha RP, McCaffrey J, O'Donnell D, Sheils O, O'Leary J, Rudman S, McDermott R, Finn S. ExPeCT: a randomised trial examining the impact of exercise on quality of life in men with metastatic prostate cancer. Support Care Cancer. 2023 Apr 22;31(5):292. doi: 10.1007/s00520-023-07740-4. PMID 37086362
- [Background] Shero ST, Benzo R, Cooper LS, Finkelstein J, Forman DE, Gaalema DE, Joseph L, Keteyian SJ, Peterson PN, Punturieri A, Zieman S, Fleg JL. Update on RFA Increasing Use of Cardiac and Pulmonary Rehabilitation in Traditional and Community Settings NIH-Funded Trials: ADDRESSING CLINICAL TRIAL CHALLENGES PRESENTED BY THE COVID-19 PANDEMIC. J Cardiopulm Rehabil Prev. 2022 Jan 1;42(1):10-14. doi: 10.1097/HCR.0000000000000635. PMID 34508036
- [Background] Siegel DA, O'Neil ME, Richards TB, Dowling NF, Weir HK. Prostate Cancer Incidence and Survival, by Stage and Race/Ethnicity - United States, 2001-2017. MMWR Morb Mortal Wkly Rep. 2020 Oct 16;69(41):1473-1480. doi: 10.15585/mmwr.mm6941a1. PMID 33056955
- [Background] Siegel RL, Miller KD, Wagle NS, Jemal A. Cancer statistics, 2023. CA Cancer J Clin. 2023 Jan;73(1):17-48. doi: 10.3322/caac.21763. PMID 36633525
- [Background] Smiley A, Tsai TY, Cui W, Parvanova I, Lyu J, Zakashansky E, Xhakli T, Cui H, Finkelstein J. Telemonitoring of Home-Based Biking Exercise: Assessment of Wireless Interfaces. JMIR Biomed Eng. 2022 Oct 12;7(2):e41782. doi: 10.2196/41782. PMID 38875588
- [Background] Smiley A, Finkelstein J. Aerobic exercise system for home telerehabilitation. 2022 IEEE 35th International Symposium on Computer-Based Medical Systems (CBMS), 2022, pp. 297-301.
- [Background] Smiley A, Tsai TY, Havrylchuk I, Cui W, Parvanova I, Zakashansky E, Xhakli T, Cui H, Finkelstein J. Development and Evaluation of Wireless Interfaces to Monitor and Control Cycling Exercise During Home Telerehabilitation. Med Devices (Auckl). 2023 Jan 19;16:1-13. doi: 10.2147/MDER.S392999. eCollection 2023. PMID 36698919
- [Background] Smiley A, Tsai TY, Zakashansky E, Gabriel A, Xhakli T, Cui W, Huo X, Havrylchuk I, Cui H, Finkelstein J. Exercise Exertion Levels Prediction Based on Real-Time Wearable Physiological Signal Monitoring. Stud Health Technol Inform. 2023 Jun 29;305:172-175. doi: 10.3233/SHTI230454. PMID 37386988
- [Background] Smith MR, Finkelstein JS, McGovern FJ, Zietman AL, Fallon MA, Schoenfeld DA, Kantoff PW. Changes in body composition during androgen deprivation therapy for prostate cancer. J Clin Endocrinol Metab. 2002 Feb;87(2):599-603. doi: 10.1210/jcem.87.2.8299. PMID 11836291
- [Background] Stacey FG, James EL, Chapman K, Courneya KS, Lubans DR. A systematic review and meta-analysis of social cognitive theory-based physical activity and/or nutrition behavior change interventions for cancer survivors. J Cancer Surviv. 2015 Jun;9(2):305-38. doi: 10.1007/s11764-014-0413-z. Epub 2014 Nov 29. PMID 25432633
- [Background] Stout NL, Santa Mina D, Lyons KD, Robb K, Silver JK. A systematic review of rehabilitation and exercise recommendations in oncology guidelines. CA Cancer J Clin. 2021 Mar;71(2):149-175. doi: 10.3322/caac.21639. Epub 2020 Oct 27. PMID 33107982
- [Background] Stone P, Hardy J, Huddart R, A'Hern R, Richards M. Fatigue in patients with prostate cancer receiving hormone therapy. Eur J Cancer. 2000 Jun;36(9):1134-41. doi: 10.1016/s0959-8049(00)00084-8. PMID 10854947
- [Background] Svynarenko R, Lindley LC. Defining Rurality in Hospice Research: Evaluation of Common Measures. J Health Care Poor Underserved. 2021;32(4):2167-2180. doi: 10.1353/hpu.2021.0189. PMID 34803066
- [Background] Sweet SN, Michalovic E, Latimer-Cheung AE, Fortier M, Noreau L, Zelaya W, Martin Ginis KA. Spinal Cord Injury Peer Mentorship: Applying Self-Determination Theory to Explain Quality of Life and Participation. Arch Phys Med Rehabil. 2018 Mar;99(3):468-476.e12. doi: 10.1016/j.apmr.2017.08.487. Epub 2017 Sep 22. PMID 28947164
- [Background] Stacey FG, James EL, Chapman K, Lubans DR. Social cognitive theory mediators of physical activity in a lifestyle program for cancer survivors and carers: findings from the ENRICH randomized controlled trial. Int J Behav Nutr Phys Act. 2016 Apr 14;13:49. doi: 10.1186/s12966-016-0372-z. PMID 27075417
- [Background] Street RL Jr, Mazor KM, Arora NK. Assessing Patient-Centered Communication in Cancer Care: Measures for Surveillance of Communication Outcomes. J Oncol Pract. 2016 Dec;12(12):1198-1202. doi: 10.1200/JOP.2016.013334. Epub 2016 Sep 30. No abstract available. PMID 27650836
- [Background] Teleni L, Chan RJ, Chan A, Isenring EA, Vela I, Inder WJ, McCarthy AL. Exercise improves quality of life in androgen deprivation therapy-treated prostate cancer: systematic review of randomised controlled trials. Endocr Relat Cancer. 2016 Feb;23(2):101-12. doi: 10.1530/ERC-15-0456. Epub 2015 Nov 19. PMID 26584972
- [Background] Thomas J, Harden A. Methods for the thematic synthesis of qualitative research in systematic reviews. BMC Med Res Methodol. 2008 Jul 10;8:45. doi: 10.1186/1471-2288-8-45. PMID 18616818
- [Background] Thompson-Leduc P, Clayman ML, Turcotte S, Legare F. Shared decision-making behaviours in health professionals: a systematic review of studies based on the Theory of Planned Behaviour. Health Expect. 2015 Oct;18(5):754-74. doi: 10.1111/hex.12176. Epub 2014 Feb 16. PMID 24528502
- [Background] Tittle MB, McMillan SC, Hagan S. Validating the brief pain inventory for use with surgical patients with cancer. Oncol Nurs Forum. 2003 Mar-Apr;30(2):325-30. doi: 10.1188/03.ONF.325-330. PMID 12692666
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- [Background] Trinh L, Plotnikoff RC, Rhodes RE, North S, Courneya KS. Feasibility and preliminary efficacy of adding behavioral counseling to supervised physical activity in kidney cancer survivors: a randomized controlled trial. Cancer Nurs. 2014 Sep-Oct;37(5):E8-22. doi: 10.1097/NCC.0b013e3182a40fb6. PMID 24232192
- [Background] Trinh L, Plotnikoff RC, Rhodes RE, North S, Courneya KS. Changes in motivational outcomes following a supervised physical activity program with behavioral counseling in kidney cancer survivors: a pilot study. Psychooncology. 2015 Sep;24(9):1204-7. doi: 10.1002/pon.3754. Epub 2015 Jan 27. No abstract available. PMID 25628184
- [Background] Tseng YF, Wang KL, Lin CY, Lin YT, Pan HC, Chang CJ. Predictors of smoking cessation in Taiwan: using the theory of planned behavior. Psychol Health Med. 2018 Mar;23(3):270-276. doi: 10.1080/13548506.2017.1378820. Epub 2017 Sep 20. PMID 28931309
- [Background] Tudge J, Mokrova I, Karnik RB, Hatfield BE. Uses and misuses of Bronfenbrenner's bioecological theory of human development. Journal of Family Theory & Review 2011;1(4):198-210.
- [Background] USDA ERS - Rural-Urban Commuting Area (RUCA) Codes. https://www.ers.usda.gov/data-products/ruralurban-commuting-area-codes/ (accessed August 21, 2023).
- [Background] Ussing A, Mikkelsen MK, Villumsen BR, Wejlgaard J, Bistrup PE, Birkefoss K, Bandholm T. Supervised exercise therapy compared with no exercise therapy to reverse debilitating effects of androgen deprivation therapy in patients with prostate cancer: a systematic review and meta-analysis. Prostate Cancer Prostatic Dis. 2022 Sep;25(3):491-506. doi: 10.1038/s41391-021-00450-0. Epub 2021 Sep 6. PMID 34489536
- [Background] Van Blarigan EL, Kenfield SA, Tantum L, Cadmus-Bertram LA, Carroll PR, Chan JM. The Fitbit One Physical Activity Tracker in Men With Prostate Cancer: Validation Study. JMIR Cancer. 2017 Apr 18;3(1):e5. doi: 10.2196/cancer.6935. PMID 28420602
- [Background] van Vugt M, de Wit M, Cleijne WH, Snoek FJ. Use of behavioral change techniques in web-based self-management programs for type 2 diabetes patients: systematic review. J Med Internet Res. 2013 Dec 13;15(12):e279. doi: 10.2196/jmir.2800. PMID 24334230
- [Background] Villumsen BR, Jorgensen MG, Frystyk J, Hordam B, Borre M. Home-based 'exergaming' was safe and significantly improved 6-min walking distance in patients with prostate cancer: a single-blinded randomised controlled trial. BJU Int. 2019 Oct;124(4):600-608. doi: 10.1111/bju.14782. Epub 2019 May 14. PMID 31012238
- [Background] Wei C, Finkelstein J. Comparison of Alexa Voice and Audio Video Interfaces for Home-Based Physical Telerehabilitation. AMIA Jt Summits Transl Sci Proc. 2022 May 23;2022:496-503. eCollection 2022. PMID 35854718
- [Background] Yabroff KR, Han X, Zhao J, Nogueira L, Jemal A. Rural Cancer Disparities in the United States: A Multilevel Framework to Improve Access to Care and Patient Outcomes. JCO Oncol Pract. 2020 Jul;16(7):409-413. doi: 10.1200/OP.20.00352. Epub 2020 Jun 23. No abstract available. PMID 32574130
- [Background] Yates P, Carter R, Cockerell R, Cowan D, Dixon C, Lal A, Newton RU, Hart N, Galvao DA, Baguley B, Denniston N, Skinner T, Couper J, Emery J, Frydenberg M, Liu WH. Evaluating a multicomponent survivorship programme for men with prostate cancer in Australia: a single cohort study. BMJ Open. 2022 Feb 2;12(2):e049802. doi: 10.1136/bmjopen-2021-049802. PMID 35110307
- [Background] Yount S, Cella D, Banik D, Ashraf T, Shevrin D. Brief assessment of priority symptoms in hormone refractory prostate cancer: the FACT Advanced Prostate Symptom Index (FAPSI). Health Qual Life Outcomes. 2003 Nov 21;1:69. doi: 10.1186/1477-7525-1-69. PMID 14633279
- [Background] Zahnd WE, James AS, Jenkins WD, Izadi SR, Fogleman AJ, Steward DE, Colditz GA, Brard L. Rural-Urban Differences in Cancer Incidence and Trends in the United States. Cancer Epidemiol Biomarkers Prev. 2018 Nov;27(11):1265-1274. doi: 10.1158/1055-9965.EPI-17-0430. Epub 2017 Jul 27. PMID 28751476
- [Background] Zahnd WE, Fogleman AJ, Jenkins WD. Rural-Urban Disparities in Stage of Diagnosis Among Cancers With Preventive Opportunities. Am J Prev Med. 2018 May;54(5):688-698. doi: 10.1016/j.amepre.2018.01.021. Epub 2018 Mar 15. PMID 29550163
- [Background] Zahnd WE, Davis MM, Rotter JS, Vanderpool RC, Perry CK, Shannon J, Ko LK, Wheeler SB, Odahowski CL, Farris PE, Eberth JM. Rural-urban differences in financial burden among cancer survivors: an analysis of a nationally representative survey. Support Care Cancer. 2019 Dec;27(12):4779-4786. doi: 10.1007/s00520-019-04742-z. Epub 2019 Apr 10. PMID 30972645
- [Background] Ziegler A. Generalized Estimating Equations. Springer, 2011. ISBN 978-1-4614-0498-9